CLINICAL TRIAL: NCT07325292
Title: A Randomized, Phase 3, Open-label Study to Investigate Pharmacokinetics, Safety, and Efficacy of Subcutaneous Compared to Intravenous Frexalimab in Adult Participants With Multiple Sclerosis
Brief Title: Non-inferiority Study of Frexalimab Subcutaneous Administration Compared to Intravenous Administration in Adult Participants With Multiple Sclerosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC18098; 2024-519304-28 (Registry Identifier: CTIS); U1111-1306-7563 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Frexalimab SC (Experimental): Frexalimab SC
  Interventions: Drug: Frexalimab; Drug: MRI contrast-enhancing preparations
- Frexalimab IV (Experimental): Frexalimab IV
  Interventions: Drug: Frexalimab; Drug: MRI contrast-enhancing preparations

INTERVENTIONS:
Drug: Frexalimab — Pharmaceutical form:Solution for injection-Route of administration:SC injection
  Other Names: SAR441344
  Arms: Frexalimab SC
Drug: Frexalimab — Pharmaceutical form:Concentrate for solution for infusion-Route of administration:IV infusion
  Other Names: SAR441344
  Arms: Frexalimab IV
Drug: MRI contrast-enhancing preparations — Route of administration:IV injection

SUMMARY:
This is a randomized, open-label, parallel, Phase 3 study with 2-arms for treatment.

The purpose of this study is to evaluate SC administration of frexalimab every 4 weeks (q4w) compared to IV administration of frexalimab q4w in male and female participants with RMS and nrSPMS (aged 18 to 60 years at the time of enrollment). People diagnosed with MS are eligible for enrollment as long as they meet all the inclusion criteria and none of the exclusion criteria.

Study details include:

The study intervention duration will be 48 weeks (12 months) for Parts A and B combined. Optional Part C will last until the initiation of a long term safety study for Frexalimab.The follow up duration after the end of study intervention (in case of discontinuation) will be 6 months.

The number of scheduled visits (Parts A and B) will be 17 or 11 for participants receiving frexalimab SC or IV, respectively, with an on-site visit frequency of every month between Week 4 and Week 24 in Part A, then every 1 to 3 months in Part B, then every 6 months in Part C. Participants discontinuing treatment before the End of Study will have an additional 3 follow-up visits.

ELIGIBILITY:
Inclusion Criteria: The participant must qualify for inclusion per either Group A or B criteria as detailed below, meeting all the inclusion criteria of the applicable group:

Group A (RMS)

* The participant must be 18 to 55 years of age, inclusive, at the time of signing the informed consent.
* The participant must have been diagnosed with RMS.
* The participant must have an Expanded Disability Status Scale (EDSS) score of ≤5.5 at the first visit (Screening Visit).
* The participant must have at least 1 of the following prior to screening:

  * 1 documented relapse within the previous year OR
  * 2 documented relapses within the previous 2 years, OR
  * 1 documented Gd enhancing lesion on an MRI scan within the previous year. Group B (nrSPMS)
* Participant must have a previous diagnosis of RRMS in accordance with the 2017 revised McDonald criteria
* The participant must be 18 to 60 years of age, inclusive, at the time of signing the informed consent.
* The participant must have a current diagnosis of SPMS.
* The participant must have documented evidence of disability progression observed during the 12 months before screening.
* The participant must have an absence of clinical relapses for at least 24 months.
* The participant must have an EDSS score between 3.0 and 6.5 points, inclusive, at the first visit (Screening Visit).

Participants from Group A and Group B are eligible to be included in the study only if all of the following criteria also apply:

- Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* The participant has been diagnosed with primary progressive MS.
* The participant has a history of infection or may be at risk for infection:
* Fever within 28 days of the Screening Visit
* Presence of psychiatric disturbance or substance abuse
* History, clinical evidence, suspicion or significant risk for thromboembolic events, as well as myocardial infarction, stroke, and/or antiphospholipid syndrome and any participants requiring antithrombotic treatment.
* Current hypogammaglobulinemia defined by Ig levels (IgG and/or IgM) below the LLN at screening or a history of primary hypogammaglobulinemia.
* A history or presence of disease that can mimic MS symptoms.
* The participant has a contraindication for MRI. The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Area under the curve over the interval W20 to W24 | Until Week 24
  AUCW20-W24
Trough concentration at steady state | Until Week 24
  Ctrough,SS

SECONDARY OUTCOMES:
Frexalimab plasma concentrations over time | Until Week 24
Pharmacokinetic parameters: Cmax | Until Week 24
Pharmacokinetic parameters: Tmax | Until Week 24
Number of participants with adverse events, SAEs, AEs leading to permanent study intervention discontinuation, AESIs, and potentially clinically significant abnormality(PCSA) in laboratory tests, and vital signs during the study period | Until Week 96
Incidence of ADAs over time | Until Week 96
Total number of Gd-enhancing T1 lesions at W12 and W24 | At Week 12 and Week 24

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Alabama Neurology Associates- Site Number : 8400115, Homewood, Alabama
  - Private Practice - Dr. Regina Berkovich- Site Number : 8400005, West Hollywood, California
  - Neurology of Central Florida- Site Number : 8400147, Altamonte Springs, Florida
  - Piedmont HealthCare - Lake Norman Neurology- Site Number : 8400002, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC18098 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=27012&tenant=MT_SNY_9011